CLINICAL TRIAL: NCT03937271
Title: Using the Objective Measurement Methods and TCM Questionnaire to Explore the Association Among TCM Pattern, TCM Tongue Diagnosis and TCM Pulse Diagnosis for Autoimmune Disease and Dry Eye Syndrome
Brief Title: Objective Measurement Methods for Autoimmune Disease and Dry Eye Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Leak of research funding
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-10-003AC
Record Dates: First submitted 2019-04-22; First posted 2019-05-03 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Sjögren's Syndrome; Systemic Lupus Erythematosus; Rheumatoid Arthritis; Systemic Sclerosis; Ankylosing Spondylitis; Dry Eye Syndrome
Keywords: Sjögren's syndrome; Systemic lupus erythematosus; Rheumatoid Arthritis; Systemic Sclerosis; Ankylosing spondylitis; Dry eye syndrome
MeSH Terms: conditions — Sjogren's Syndrome; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Scleroderma, Systemic; Spondylitis, Ankylosing; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Sjögren's syndrome: Sjögren's syndrome patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 2002 American-European Consensus Criteria for SS (AECG)
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test
- Systemic lupus erythematosus: Systemic lupus erythematosus patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 1982 revised Systemic lupus erythematosus criteria
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test
- Rheumatoid Arthritis: Rheumatoid Arthritis patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 2010 ACR/EULAR Rheumatoid Arthritis classification criteria
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test
- Systemic Sclerosis: Systemic Sclerosis patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 1980 ACR eSystemic Sclerosis criteria
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test
- Ankylosing spondylitis: Ankylosing spondylitis patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) fulfilled the 1984 Ankylosing spondylitis Modified New York criteria
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test
- Dry eye syndrome: Dry eye syndrome patients were screened in the ophthalmology outpatient departments, rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 20 and 75 years; (2) Schirmer's test less than 10 mm/5 min
  Interventions: Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test

INTERVENTIONS:
Diagnostic Test: Traditional Chinese Medicine pattern — Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS) for comparing with the Dry eye syndrome (DES) subjects will take the Traditional Chinese Medicine pattern.
Diagnostic Test: Traditional Chinese Medicine tongue diagnosis — Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS) for comparing with the Dry eye syndrome (DES) subjects will take the Traditional Chinese Medicine tongue diagnosis.
Diagnostic Test: Traditional Chinese Medicine pulse diagnosis — Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS) for comparing with the Dry eye syndrome (DES) subjects will take the Traditional Chinese Medicine pulse diagnosis.
Diagnostic Test: Heart rate variability — Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS) for comparing with the Dry eye syndrome (DES) subjects will take the Heart rate variability.
Diagnostic Test: Schirmer's test — Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS) for comparing with the Dry eye syndrome (DES) subjects will take the Schirmer's test.

SUMMARY:
To explore the association among TCM pattern, TCM tongue diagnosis and TCM pulse diagnosis for Autoimmune disease and Dry eye syndrome

DETAILED DESCRIPTION:
Objective: To explore the association among TCM pattern, TCM tongue diagnosis and TCM pulse diagnosis for Autoimmune disease and Dry eye syndrome

Method:

This study wants to establish the objective measurement of Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS) for comparing with the Dry eye syndrome (DES) subjects. And the investigators want to use the objective measurement tools to explore the association of TCM pattern, heart rate variability (HRV), TCM tongue diagnosis and TCM pulse diagnosis among at least 50 each AID group subjects and at least 50 DES subjects.

Expected Results:

1. To evaluate the difference among TCM pattern, HRV, TCM tongue diagnosis, TCM pulse diagnosis for the each AID groups.
2. To evaluate the difference among TCM pattern, HRV, TCM tongue diagnosis, TCM pulse diagnosis for the each DES groups.
3. To evaluate the difference among TCM pattern, HRV, TCM tongue diagnosis, TCM pulse diagnosis among the AID groups and DES group.

Keyword: Autoimmune disease, Dry eye syndrome, TCM pattern, TCM tongue diagnosis, TCM pulse diagnosis

ELIGIBILITY:
Sjögren's syndrome

Inclusion Criteria:

* (1) aged between 20 and 75 years
* (2) fulfilled the 2002 American-European Consensus Criteria for SS (AECG) Exclusion Criteria: NA

Systemic lupus erythematosus

Inclusion Criteria:

* (1) aged between 20 and 75 years
* (2) fulfilled the 1982 ACR revised Systemic lupus erythematosus criteria Exclusion Criteria: NA

Rheumatoid Arthritis

Inclusion Criteria:

* (1) aged between 20 and 75 years
* (2) fulfilled the 2010 ACR/EULAR Rheumatoid Arthritis classification criteria Exclusion Criteria: NA

Systemic Sclerosis

Inclusion Criteria:

* (1) aged between 20 and 75 years
* (2) fulfilled the 1980 ACR eSystemic Sclerosis criteria Exclusion Criteria: NA

Ankylosing spondylitis

Inclusion Criteria:

* (1) aged between 20 and 75 years
* (2) fulfilled the 1984 Ankylosing spondylitis Modified New York criteria Exclusion Criteria: NA

Dry eye syndrome

Inclusion Criteria:

* (1) aged between 20 and 75 years
* (2) Schirmer's test less than 10 mm/5 min

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Autoimmune disease (AID) as Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS), and Dry eye syndrome (DES) subjects were screened in the ophthalmology outpatient departments, rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
TCM pattern | Five year
  TCM pattern is a tool for detecting the constitution among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS), and Dry eye syndrome (DES).
TCM tongue diagnosis | Five year
  TCM tongue diagnosis is a tool for detecting tongue expression among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS), and Dry eye syndrome (DES).
TCM pulse diagnosis | Five year
  TCM pulse diagnosis is a tool for detecting pulse of radial artery among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS), and Dry eye syndrome (DES) .
Heart rate variability (HRV) | Five year
  HRV is a tool for detecting the ratio between High-frequency (HF) activity and low-frequency (LF) activity. among the Sjögren's syndrome (SJS), Systemic lupus erythematosus (SLE), Rheumatoid Arthritis (RA), Systemic Sclerosis (SSc), Ankylosing spondylitis (AS), and Dry eye syndrome (DES) .

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Mao Chang, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Ching-Mao Chang, Taipei, Taiwan (r.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No